CLINICAL TRIAL: NCT05715437
Title: Analgesic Efficacy of Adductor Canal Block With Bupivacaine Versus Bupivacaine and Ketamine in Total Knee Arthroplasty.
Brief Title: Adductor Canal Block in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ehab William Samir, Principal Investigator, Assiut University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: Adductor canal block
Record Dates: First submitted 2023-01-23; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Saline Solution; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine plus Normal Saline (Experimental): 30 patients will receive bolus shot 20ml of 0.5% of Bupivacaine plus 1ml Normal saline postoperative TKA.
  Interventions: Drug: Bupivacaine plus Normal Saline
- Bupivacaine and Ketamine (Experimental): 30 patients will receive bolus shot 20ml of 0.5% of Bupivacaine plus 1ml ketamine (50mg) postoperative TKA.
  Interventions: Drug: Bupivacain and ketamine

INTERVENTIONS:
Drug: Bupivacaine plus Normal Saline — Effect of Bupivacain and ketamine and is superior to Bupivacaine and Normal Saline in terms of providing better pain control for 48 hours postoperatively after TKA.
  Arms: Bupivacaine plus Normal Saline
Drug: Bupivacain and ketamine — Effect of Bupivacain and ketamine and is superior to Bupivacaine and Normal Saline in terms of providing better pain control for 48 hours postoperatively after TKA.
  Arms: Bupivacaine and Ketamine

SUMMARY:
The purpose of this study is to evaluate whether adding ketamine to bupivacaine is superior to bupivacaine alone in terms of providing better pain control for 48 hours postoperatively after TKA.

DETAILED DESCRIPTION:
Optimal pain relief is essential for functional recovery after total knee arthroplasty (TKA). Addition of femoral nerve block (FNB) to an analgesic regimen provides superior pain control and shortens hospital stay, in comparison with epidural or intravenous patient-controlled analgesia (PCA) alone. However, prolonged motor blockade from FNB is associated with a small (2%) but clinically important risk of fall. With FNB there will always be a compromise between the goals of adequate pain relief and muscle strength. An ideal nerve block would provide effective analgesia, minimize opioid use and side effects, and hasten mobilization by preserving motor strength. "Fast-track" total joint replacements are gaining popularity. Motor preservation with adequate analgesia has become the optimal postoperative pain goal in orthopedic surgeries to enable earlier physical therapy, faster recovery, and shorter hospital stays.Nerve blocks such as femoral nerve block, adductor canal block, and epidural block have been more prevalent in TKA postoperative analgesia due to their effectiveness, easy manipulation, and low rate of complications. Local anesthetics such as ropivacaine or bupivacaine have been commonly used in nerve blocks. However, the postoperative analgesic effects and duration of local anesthetics are not good enough, and sometimes have led to delayed ambulation and an increased risk of falling after TKA. To overcome these shortcomings and further improve the analgesic effect, additional endeavors should be devoted to exploring new and effective agents for nerve block.With the advent of ultrasonography, the adductor canal can be easily visualized at the mid-thigh level, allowing performance of adductor canal block (ACB) with a high success rate. In recent years, ACB has been successfully used for postoperative pain control after knee surgery. Anatomical study of the adductor canal demonstrated that the adductor canal may serve as a conduit for more than just the saphenous nerve, possibly including the vastus medialis nerve, medial femoral cutaneous nerve, articular branches from the obturator nerve, as well as the medial retinacular nerve. Thus, the sensory changes are not limited to the distribution of the saphenous nerve, but includes the medial and anterior aspects of the knee from the superior pole of the patella to the proximal tibia.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is scheduled for elective primary unilateral TKA.
2. The subject is ≥ 18 years and ≤ 80 years.
3. Both sexes.
4. The subject's primary anesthesia care team has planned for a spinal anesthesia.
5. The patient agrees to receive an adductor canal block.
6. ASA class 1-3.

Exclusion Criteria:

1. Subject is < 18 years of age or >80 years of age.
2. Subject is known or believed to be pregnant.
3. Significant pre-existing neuropathy on the operative limb.
4. Significant renal, cardiac or hepatic disease.
5. ASA class 4-5.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 48 hours
  Maximum postoperative pain assessment by the visual analogue scale (VAS) pain scores in the first 48 hours.

SECONDARY OUTCOMES:
analgesia | 48 hours
  VAS pain scores when the knee joint was bent to 45°. At 4 ,8,12,24,36 and 48 hours.
Analysis include quadriceps strength | 48 hours
  quadriceps strength, each of which were assessed at 4, 24, and 48 hours after the operation. The following 5-grade scale was used to quantify quadriceps strength: 1=could not contract; 2=could contract, but the contraction could not cause the knee joint to move; 3=could bear gravity, but could not bear any substantial resistance; 4=could bear substantial resistance; 5=could bear full resistance.
Satisfaction of the patients | 48 hours
  measured using "Likert scale" was acceptable (very satisfied, satisfied, neutral)
Reporting side effects of drugs given | 48 hours
  Side effects of Ketamine: tachycardia, increase blood pressure , allergic reaction, confusion , delirium , hallucination and nightmares.
  Side effects of Bupivacaine: chest pain and discomfort, difficult breathing, muscle stiffness, abnormal heart rhythms, numbness or tingling around your mouth, and allergic reaction.

REFERENCES:
- [Background] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Background] Allen HW, Liu SS, Ware PD, Nairn CS, Owens BD. Peripheral nerve blocks improve analgesia after total knee replacement surgery. Anesth Analg. 1998 Jul;87(1):93-7. doi: 10.1097/00000539-199807000-00020. PMID 9661553
- [Background] Hadzic A, Houle TT, Capdevila X, Ilfeld BM. Femoral nerve block for analgesia in patients having knee arthroplasty. Anesthesiology. 2010 Nov;113(5):1014-5. doi: 10.1097/ALN.0b013e3181f4b43d. No abstract available. PMID 20881593
- [Background] Wang H, Boctor B, Verner J. The effect of single-injection femoral nerve block on rehabilitation and length of hospital stay after total knee replacement. Reg Anesth Pain Med. 2002 Mar-Apr;27(2):139-44. doi: 10.1053/rapm.2002.29253. PMID 11915059
- [Background] Singelyn FJ, Deyaert M, Joris D, Pendeville E, Gouverneur JM. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous three-in-one block on postoperative pain and knee rehabilitation after unilateral total knee arthroplasty. Anesth Analg. 1998 Jul;87(1):88-92. doi: 10.1097/00000539-199807000-00019. PMID 9661552
- [Background] YaDeau JT, Cahill JB, Zawadsky MW, Sharrock NE, Bottner F, Morelli CM, Kahn RL, Sculco TP. The effects of femoral nerve blockade in conjunction with epidural analgesia after total knee arthroplasty. Anesth Analg. 2005 Sep;101(3):891-895. doi: 10.1213/01.ANE.0000159150.79908.21. PMID 16116010